CLINICAL TRIAL: NCT01197755
Title: (OSKIRA-3): A Phase III, Multi-centre, Randomised, Double-Blind, Placebo-Controlled, Parallel Group Study of Two Dosing Regimens of Fostamatinib Disodium in Rheumatoid Arthritis Patients With Inadequate Response to a TNF-alpha Antagonist
Brief Title: Evaluation of Effectiveness of Two Dosing Regimens of Fostamatinib Compared to Placebo in Patients With Rheumatoid Arthritis (RA) Who Are Taking Methotrexate and Have Had Inadequate Response to Single TNF-alpha Antagonist
Acronym: OSKIRA - 3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D4300C00003; 2010-020745-27 (EudraCT Number)
Record Dates: First submitted 2010-09-08; First posted 2010-09-09 (Estimated); Results first posted 2014-04-07 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — fostamatinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dosing Regimen A (Experimental): Oral Treatment
  Interventions: Drug: fostamatinib
- Dosing Regimen B (Experimental): Oral Treatment
  Interventions: Drug: fostamatinib
- Dosing Regimen C (Placebo Comparator): Oral Treatment
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: fostamatinib — fostamatinib 100 mg twice daily
  Arms: Dosing Regimen A
Drug: fostamatinib — fostamatinib 100 mg twice daily/150 mg once daily
  Arms: Dosing Regimen B
Drug: placebo — Placebo twice daily
  Arms: Dosing Regimen C

SUMMARY:
The purpose of the study is to evaluate the effectiveness of two dosing regimens of fostamatinib compared to placebo, in patients with rheumatoid arthritis (RA) who are taking methotrexate and have had an inadequate response to a single TNF-alpha antagonist. The study will last for approximately six months.

DETAILED DESCRIPTION:
Sub-study:

Full title: Optional Genetic Research

Date: 18 June 2010

Version: 1

Objectives: To collect and store, with appropriate consent ,DNA samples for future exploratory research into genes/genetic variation that may influence response (ie, absorption, distribution, metabolism and excretion, safety, tolerability and efficacy) to fostamatinib disodium and/or methotrexate; and/or susceptibility to, progression of and prognosis of RA

ELIGIBILITY:
Inclusion Criteria:

* Active rheumatoid arthritis (RA) diagnosed after the age of 16
* Currently taking methotrexate
* 6 or more swollen joints and 6 or more tender/painful joints (from 28 joint count) and either Erythrocyte Sedimentation Rate (ESR) blood result of 28mm/h or more, or C-Reactive Protein (CRP) blood result of 10mg/L or more
* At least one of the following: documented history of positive rheumatoid factor (blood test), current presence of rheumatoid factor (blood test), radiographic erosion within 12months prior to study enrolment, presence of serum anti-cyclic citrullinated peptide antibodies (blood test)

Exclusion Criteria:

* Females who are pregnant or breast feeding
* Poorly controlled hypertension
* Liver disease or significant liver function test abnormalities
* Certain inflammatory conditions (other than rheumatoid arthritis), connective tissue diseases or chronic pain disorders
* Recent or significant cardiovascular disease
* Significant active or recent infection including tuberculosis
* Previous failure to respond to anakinra or previous treatment with biological agent (other than TNF alpha antagonists including rituximab, abatacept and tocilizumab)
* Severe renal impairment
* Neutropenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2010-09; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil MacKillop, MD PhD, Study Director — AstraZeneca
Locations (135):
- United States (67):
  - Research Site, Anniston, Alabama
  - Research Site, Huntsville, Alabama
  - Research Site, Tuscaloosa, Alabama
  - Research Site, Mesa, Arizona
  - Research Site, Scottsdale, Arizona
  - Research Site, Hot Springs, Arkansas
  - Research Site, Glendale, California
  - Research Site, La Jolla, California
  - Research Site, Long Beach, California
  - Research Site, Palo Alto, California
  - Research Site, Santa Maria, California
  - Research Site, Torrance, California
  - Research Site, Tustin, California
  - Research Site, Upland, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, Bridgeport, Connecticut
  - Research Site, Trumbull, Connecticut
  - Research Site, Lewes, Delaware
  - Research Site, Brandon, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Ocala, Florida
  - Research Site, Orlando, Florida
  - Research Site, Tampa, Florida
  - Research Site, Venice, Florida
  - Research Site, Zephyrhills, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Canton, Georgia
  - Research Site, Idaho Falls, Idaho
  - Research Site, Decatur, Illinois
  - Research Site, Cedar Rapids, Iowa
  - Research Site, Bowling Green, Kentucky
  - Research Site, Elizabethtown, Kentucky
  - Research Site, Crofton, Maryland
  - Research Site, Fall River, Massachusetts
  - Research Site, Worcester, Massachusetts
  - Research Site, Lansing, Michigan
  - Research Site, Flowood, Mississippi
  - Research Site, Florissant, Missouri
  - Research Site, Richmond Heights, Missouri
  - Research Site, Las Cruces, New Mexico
  - Research Site, Albany, New York
  - Research Site, Brooklyn, New York
  - Research Site, Olean, New York
  - Research Site, Rochester, New York
  - Research Site, Roslyn, New York
  - Research Site, Smithtown, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, Dayton, Ohio
  - Research Site, Mayfield Village, Ohio
  - Research Site, Lake Oswego, Oregon
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, West Reading, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Greenville, South Carolina
  - Research Site, Hixson, Tennessee
  - Research Site, Memphis, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Amarillo, Texas
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Tacoma, Washington
- Argentina (10):
  - Research Site, Buenos Aires, Buenos Aires F.D.
  - Research Site, Córdoba, CRD
  - Research Site, Rosario, Santa Fe Province
  - Research Site, San Miguel de Tucumán, TUC
  - Research Site, Buenos Aires
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Quilmes
  - Research Site, Rosario
  - Research Site, San Juan
  - Research Site, San Miguel de Tucumán
- Belgium (4):
  - Research Site, Brussels, Belgium
  - Research Site, Ghent, Belgium
  - Research Site, Liège, Belgium
  - Research Site, Yvoir
- Brazil (4):
  - Research Site, Porto Alegre, Brasil
  - Research Site, Goiânia, Goiás
  - Research Site, Curitiba, Paraná
  - Research Site, São Paulo, São Paulo
- Canada (5):
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Mississauga, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Pointe-Claire, Quebec
  - Research Site, Rimouski, Quebec
- Czechia (6):
  - Research Site, Bruntál
  - Research Site, České Budějovice
  - Research Site, Hlučín
  - Research Site, Ostrava-trebovice
  - Research Site, Prague
  - Research Site, Zlín
- Research Site, Orléans, France
- Germany (8):
  - Research Site, Hamburg, Hamburg
  - Research Site, Aachen, North Rhine-Westphalia
  - Research Site, Leipzig, Saxony
  - Research Site, Erlangen
  - Research Site, Frankfurt
  - Research Site, Hamburg
  - Research Site, Heidelberg
  - Research Site, München
- Research Site, Budapest, Hungary
- Israel (5):
  - Research Site, Ashkelon
  - Research Site, Haifa
  - Research Site, Kfar Saba
  - Research Site, Ramat Gan
  - Research Site, Tel Litwinsky
- Italy (2):
  - Research Site, Iesi, AN
  - Research Site, Ferrara, FE
- Mexico (5):
  - Research Site, Chihuahua City, Chihuahua
  - Research Site, Obrergon, Sonora
  - Research Site, DF
  - Research Site, Monterrey
  - Research Site, Saltillo
- Portugal (2):
  - Research Site, Lisbon
  - Research Site, Porto
- South Africa (3):
  - Research Site, Cape Town
  - Research Site, Pretoria
  - Research Site, Stellenbosch
- Research Site, Barcelona, Spain
- United Kingdom (11):
  - Research Site, Reading, Berkshire
  - Research Site, Warrington, Cheshire
  - Research Site, Maidstone, Kent
  - Research Site, Eastbourne, Sussex
  - Research Site, Cambridge
  - Research Site, Christchurch
  - Research Site, Ipswich
  - Research Site, London
  - Research Site, Metropolitan Borough of Wirral
  - Research Site, Nottingham
  - Research Site, Westcliff-on-the Sea

REFERENCES:
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=419&filename=CSR-D8480C00030.pdf
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=1201&filename=CSR-D1700C00001.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 638 patients were enrolled: 105, 108 & 110 were randomised to Groups A, B & C respectively (105, 108 & 109 received at least 1 dose of investigational product).
Pre-assignment Details: A total of 315 patients failed screening.
Groups:
- FOSTA 100 MG BID PO: Dosing Group A
- FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO: Dosing Group B
- PLACEBO PO: Dosing Group C
Period: Overall Study
Arm/Group | FOSTA 100 MG BID PO | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO | PLACEBO PO
Started | 105 (Patients who received treatment) | 108 (Patients who received treatment) | 109 (Patients who received treatment)
Randomised But Did Not Receive Treatment | 0 | 0 | 1 (Severe non-compliance to the protocol)
Completed | 67 (Number of patients who completed treatment includes patients who had a dose reduction.) | 65 (Number of patients who completed treatment includes patients who had a dose reduction.) | 55 (Number of patients who completed treatment includes patients who had a dose reduction.)
Not Completed | 38 | 43 | 54
Not completed — Adverse Event | 8 | 10 | 10
Not completed — Study-specific discontinuation criteria | 2 | 1 | 0
Not completed — Entered the long-term extension study | 18 | 21 | 35
Not completed — Lack of therapeutic response | 0 | 7 | 4
Not completed — Severe non-compliance to the protocol | 2 | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — eg, change in circumstances | 7 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FOSTA 100 MG BID PO | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO | PLACEBO PO | Total
Number analyzed (Participants) | 105 | 108 | 109 | 322
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (11.9) | 51 (12.0) | 53 (13.0) | 53 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 87 | 85 | 261
  Male | 16 | 21 | 24 | 61
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 86 | 92 | 91 | 269
  Black or African American | 9 | 5 | 9 | 23
  Asian | 0 | 1 | 0 | 1
  American Indian or Alaska Native | 1 | 4 | 1 | 6
  Indian or Pakistani | 2 | 0 | 1 | 3
  Other | 7 | 6 | 7 | 20

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Achieving ACR20 at Week 24, Comparison Between Fostamatinib and Placebo
Description: ACR20: American College of Rheumatology 20% response criteria, based on count of swollen and tender joints (out of 28 joints), blood test measures of inflammation (such as C-Reactive Protein) and the physician and patient's own assessments of disease activity, pain and physical function. BID = twice daily, DMARD = disease-modifying anti-rheumatic drug, PO = orally, QD = once daily.
Time Frame: 24 weeks
Population: The full analysis set includes those patients who received at least 1 dose of investigational product. Patients were analysed by randomised treatment in accordance with the intention to treat principle.
Measure: Number; unit: Percentage of responders
Arm/Group | FOSTA 100 MG BID PO | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO | PLACEBO PO
Number analyzed (Participants) | 105 | 108 | 109
Percentage of responders | 36.2 | 27.8 | 21.1
Statistical Analysis 1: Comparison: FOSTA 100 MG BID PO vs PLACEBO PO; Non-responder imputation has been applied following premature withdrawal, or increased dose of methotrexate or any DMARD initiation, or for 8 weeks following receipt of any parenteral steroids, or for patients with no post baseline data; Test type: Superiority or Other; p = 0.004, Mantel Haenszel — Week 24; Treatment difference in proportion of responders at Week 24 with a Mantel-Haenszel approach stratified by pooled country; Weighted difference in proportion = 0.17, 95% CI 2-sided [0.05 to 0.28]
Statistical Analysis 2: Comparison: FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO vs PLACEBO PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.168, Mantel Haenszel — Week 24; [statistical method as in outcome 1, analysis 1]; Weighted difference in proportion = 0.07, 95% CI 2-sided [-0.03 to 0.18]

2. Secondary Outcome: Proportion of Patients Achieving ACR20 at Week 1, Comparison Between Fostamatinib and Placebo
Description: as for outcome 1
Time Frame: 1 week
Population: as for outcome 1
Measure: Number; unit: Percentage of responders
Groups:
- Dosing Group A and B Combined PO: Fostamatinib 100 mg BID (combined)
Arm/Group | PLACEBO PO | Dosing Group A and B Combined PO
Number analyzed (Participants) | 109 | 213
Percentage of responders | 3.7 | 25.4
Statistical Analysis 1: Comparison: PLACEBO PO vs Dosing Group A and B Combined PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Mantel Haenszel; 95% confidence intervals and p-values are calculated using a Mantel-Haenszel approach stratified by pooled country; Weighted difference in proportion = 0.22, 95% CI 2-sided [0.16 to 0.29]

3. Secondary Outcome: Proportion of Patients Achieving ACR50 at Week 24, Comparison Between Fostamatinib and Placebo
Description: ACR50: American College of Rheumatology 50% response criteria, based on count of swollen and tender joints (out of 28 joints), blood test measures of inflammation (such as C-Reactive Protein) and the physician and patient's own assessments of disease activity, pain and physical function. BID = twice daily, DMARD = disease-modifying anti-rheumatic drug, PO = orally, QD = once daily.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of responders
Arm/Group | FOSTA 100 MG BID PO | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO | PLACEBO PO
Number analyzed (Participants) | 105 | 108 | 109
Percentage of responders | 18.1 | 13.0 | 8.3
Statistical Analysis 1: Comparison: FOSTA 100 MG BID PO vs PLACEBO PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.014, Mantel Haenszel; 95% confidence intervals and p-values are calculated using a Mantel-Haenszel approach stratified by pooled country; Weighted difference in proportion = 0.10, 95% CI 2-sided [0.02 to 0.19]
Statistical Analysis 2: Comparison: FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO vs PLACEBO PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.180, Mantel Haenszel — Nominal p-value presented for Group B comparison. Formal statistical testing could not be carried out due to the predefined multiplicity procedure (primary variable comparison of Group B versus Group C was non-significant); 95% confidence intervals and p-values are calculated using a Mantel-Haenszel approach stratified by pooled country; Weighted difference in proportion = 0.05, 95% CI 2-sided [-0.02 to 0.12]

4. Secondary Outcome: Proportion of Patients Achieving ACR70 at Week 24, Comparison Between Fostamatinib and Placebo
Description: ACR70: American College of Rheumatology 70% response criteria, based on count of swollen and tender joints (out of 28 joints), blood test measures of inflammation (such as C-Reactive Protein) and the physician and patient's own assessments of disease activity, pain and physical function. BID = twice daily, DMARD = disease-modifying anti-rheumatic drug, PO = orally, QD = once daily.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of responders
Arm/Group | FOSTA 100 MG BID PO | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO | PLACEBO PO
Number analyzed (Participants) | 105 | 108 | 109
Percentage of responders | 14.3 | 2.8 | 2.8
Statistical Analysis 1: Comparison: FOSTA 100 MG BID PO vs PLACEBO PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Mantel Haenszel; 95% confidence intervals and p-values are calculated using a Mantel-Haenszel approach stratified by pooled country; Weighted difference in proportion = 0.12, 95% CI 2-sided [0.06 to 0.19]
Statistical Analysis 2: Comparison: FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO vs PLACEBO PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.891, Mantel Haenszel — [p-value comment as in outcome 3, analysis 2]; 95% confidence intervals and p-values are calculated using a Mantel-Haenszel approach stratified by pooled country; Weighted difference in proportion = 0.00, 95% CI 2-sided [-0.04 to 0.04]

5. Secondary Outcome: ACRn - Comparison Between Fostamatinib and Placebo at Week 24
Description: ACRn: American College of Rheumatology index of RA improvement, based on smallest percentage improvement in the count of swollen joints (out of 28 joints), count of tender joints (out of 28 joints), or in blood test measures of inflammation (such as C-Reactive Protein) or the physician or patient's own assessments of disease activity, pain and physical function. Scores are reported as a percentage improvement on a scale of -100 to +100, with larger values representing a better clinical outcome. Mean refers to change at Week 24. BID = twice daily, DMARD = disease-modifying anti-rheumatic drug, PO = orally, QD = once a day.
Time Frame: Baseline and 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage improvement from baseline
Arm/Group | FOSTA 100 MG BID PO | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO | PLACEBO PO
Number analyzed (Participants) | 105 | 108 | 109
Percentage improvement from baseline | 16.25 (36.994) | 13.00 (24.718) | 5.87 (26.726)
Statistical Analysis 1: Comparison: FOSTA 100 MG BID PO vs PLACEBO PO; Non-responder imputation has been applied following premature withdrawal, or any DMARD initiation, or for 8 weeks following receipt of any parenteral steroids, or for patients with no post baseline data; Test type: Superiority or Other; p = 0.010, Van Elteren — Nominal p-value presented for treatment comparison. ACRn was not formally tested within the predefined multiplicity procedure. As this is a non-parametric test p-values alone are presented rather than an estimated treatment difference; P-values are estimated using the Van Elteren test stratified by pooled country; Treatment difference
Statistical Analysis 2: Comparison: FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO vs PLACEBO PO; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.019, Van Elteren — [p-value comment as in outcome 5, analysis 1]; P-values are estimated using the Van Elteren test stratified by pooled country

6. Secondary Outcome: Proportion of Patients Achieving DAS28-CRP <2.6 at Week 24, Comparison Between Fostamatinib and Placebo
Description: DAS28-CRP: Disease Activity Score based on a count of swollen and tender joints (out of 28 joints), blood test measures of inflammation (CRP) and the patients' own assessment. Scores can take any positive value with a lower value indicating a better clinical condition. A DAS28-CRP score of <2.6 is indicative of remission of RA symptoms. BID = twice daily, CRP = C-reactive protein, DMARD = disease-modifying anti-rheumatic drug, OR = odds ratio, PO = orally, QD = once daily.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of responders
Arm/Group | FOSTA 100 MG BID PO | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO | PLACEBO PO
Number analyzed (Participants) | 105 | 108 | 109
Percentage of responders | 11.4 | 7.4 | 3.7
Statistical Analysis 1: Comparison: FOSTA 100 MG BID PO vs PLACEBO PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.023, Regression, Logistic; Odds ratio and 95% confidence intervals are calculated using Logistic Regression with treatment and pooled country as factors; Odds Ratio (OR) = 4.1, 95% CI 2-sided [1.21 to 13.91] — An odds ratio of >1 indicates a benefit towards fostamatinib
Statistical Analysis 2: Comparison: FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO vs PLACEBO PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.197, Regression, Logistic — [p-value comment as in outcome 3, analysis 2]; [statistical method as in outcome 6, analysis 1]; Odds Ratio (OR) = 2.3, 95% CI 2-sided [0.65 to 8.23] — An odds ratio of >1 indicates a benefit towards fostamatinib

7. Secondary Outcome: Proportion of Patients Achieving DAS28-CRP <=3.2 at Week 12, Comparison Between Fostamatinib and Placebo
Description: DAS28-CRP: Disease Activity Score based on a count of swollen and tender joints (out of 28 joints), blood test measures of inflammation (CRP) and the patients' own assessment. Scores can take any positive value with a lower value indicating a better clinical condition. A DAS28-CRP score of <=3.2 indicates low disease activity. BID = twice daily, CRP = C-reactive protein, DMARD = disease-modifying anti-rheumatic drug, OR = odds ratio, PO = orally, QD = once daily.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of responders
Arm/Group | FOSTA 100 MG BID PO | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO | PLACEBO PO
Number analyzed (Participants) | 105 | 108 | 109
Percentage of responders | 18.1 | 20.4 | 5.5
Statistical Analysis 1: Comparison: FOSTA 100 MG BID PO vs PLACEBO PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.005, Regression, Logistic; [statistical method as in outcome 6, analysis 1]; Odds Ratio (OR) = 4.1, 95% CI 2-sided [1.54 to 10.92] — An odds ratio of >1 indicates a benefit towards fostamatinib
Statistical Analysis 2: Comparison: FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO vs PLACEBO PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.002, Regression, Logistic — [p-value comment as in outcome 3, analysis 2]; [statistical method as in outcome 6, analysis 1]; Odds Ratio (OR) = 4.7, 95% CI 2-sided [1.79 to 12.30] — An odds ratio of >1 indicates a benefit towards fostamatinib

8. Secondary Outcome: Proportion of Patients Achieving DAS28-CRP EULAR Response at Week 24, Comparison Between Fostamatinib and Placebo
Description: Change from baseline in DAS28-CRP at Week 24 was categorised using the European League Against Rheumatism (EULAR) response criteria. BID = twice daily, CRP = C-reactive protein, DAS28 = Disease Activity Score based on a 28-joint count, DMARD = disease-modifying anti-rheumatic drug, OR = odds ratio, PO = orally, QD = once a day.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of responders
Arm/Group | FOSTA 100 MG BID PO | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO | PLACEBO PO
Number analyzed (Participants) | 105 | 108 | 109
Percentage of responders
  No response | 46.7 (1.46) [0.20 to 0.68] | 54.6 (1.34) [0.26 to 0.89] | 67.9 (1.30) [0.20 to 0.65]
  Moderate response | 29.5 | 34.3 | 26.6
  Good response | 23.8 | 11.1 | 5.5
Statistical Analysis 1: Comparison: FOSTA 100 MG BID PO vs PLACEBO PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Proportional odds model — Nominal p value only. This was not included in the pre-defined multiplicity testing procedure; No response, moderate response and good response are included in the proportional odds model with treatment and pooled country as factors; Odds Ratio (OR) = 3.27, 95% CI 2-sided [1.86 to 5.76] — An odds ratio >1 indicates a benefit towards fostamatinib
Statistical Analysis 2: Comparison: FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO vs PLACEBO PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.028, Proportional odds model — Nominal p-value only. This was not included in the pre-defined multiplicity testing procedure; [statistical method as in outcome 8, analysis 1]; Odds Ratio (OR) = 1.89, 95% CI 2-sided [1.07 to 3.31] — An odds ratio >1 indicates a benefit towards fostamatinib

9. Secondary Outcome: Proportion of Patients With a HAQ-DI Response at Week 24 - Comparison Between Fostamatinib and Placebo
Description: HAQ-DI: Health Assessment Questionnaire - Disability Index, a measure of physical function. The HAQ-DI score is calculated by summing the category scores from 8 sub-categories (ie, scores for patient ability in dressing and grooming, rising, eating, walking, hygeine, reach, grip and common daily activities) and dividing by the number of categories completed. The HAQ-DI score takes values between 0 and 3, with a higher score indicating greater disability. A HAQ-DI response is a reduction from baseline in HAQ-DI greater than or equal to the minimally important difference (0.22). BID = twice daily, DMARD = disease-modifying anti-rheumatic drug, OR = odds ratio, PO = orally, QD = once a day.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of responders
Arm/Group | FOSTA 100 MG BID PO | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO | PLACEBO PO
Number analyzed (Participants) | 105 | 108 | 109
Percentage of responders | 41.9 | 31.5 | 23.9
Statistical Analysis 1: Comparison: FOSTA 100 MG BID PO vs PLACEBO PO; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.004, Regression, Logistic; [statistical method as in outcome 6, analysis 1]; Odds Ratio (OR) = 2.4, 95% CI 2-sided [1.33 to 4.45] — An odds ratio >1 indicates a benefit towards fostamatinib
Statistical Analysis 2: Comparison: FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO vs PLACEBO PO; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.186, Regression, Logistic — [p-value comment as in outcome 3, analysis 2]; [statistical method as in outcome 6, analysis 1]; Odds Ratio (OR) = 1.5, 95% CI 2-sided [0.82 to 2.79] — An odds ratio >1 indicates a benefit towards fostamatinib

10. Secondary Outcome: Change From Baseline to Week 24 in mTSS Score, Comparison Between Fostamatinib and Placebo
Description: mTSS: modified total sharp score, a measure of structural progression based upon X-rays. Hand and foot joints are scored for eroisions and joint space narrowing and the results summed to give a value between 0 and 488. A higher value represents more serious progression of the disease. After disregarding ineligible records, patients with 2 or more non-missing values had missing data imputed via linear extrapolation/interpolation methods. Patients with only 1 result were excluded from the analysis. ANCOVA = Analysis of covariance, BID = twice daily, IP = investigational product, PO = orally, QD = once a day.
Time Frame: Baseline and 24 weeks
Population: The full analysis set includes patients who received at least 1 dose of IP. Patients were analysed by randomised treatment in accordance with the intention to treat principle. Measurements at 2 timepoints are required for a patient to be included in the analysis; therefore patients with only 1 result have been excluded from the analysis population.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | FOSTA 100 MG BID PO | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO | PLACEBO PO
Number analyzed (Participants) | 81 | 87 | 88
Units on a scale | 0.80 (2.636) | 0.18 (3.455) | 0.84 (1.989)
Statistical Analysis 1: Comparison: FOSTA 100 MG BID PO vs PLACEBO PO; Test type: Superiority or Other; p = 0.729, ANCOVA — Nominal p-value only. This was not included in the pre-defined multiplicity procedure. As this is a non-parametric test p-values alone are presented rather than an estimated treatment difference; This was performed on the ranks of the change from baseline, by pooled country, including a term for the ranks of the baseline score as covariate
Statistical Analysis 2: Comparison: FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO vs PLACEBO PO; Test type: Superiority or Other; p = 0.019, ANCOVA — [p-value comment as in outcome 10, analysis 1]; [statistical method as in outcome 10, analysis 1]

11. Secondary Outcome: SF-36 - Comparison of the Change in PCS From Baseline Between Fostamatinib and Placebo at Week 24
Description: SF-36: 36 item short form health survey, as a measure of health-related quality of life. Scores for 8 sub-domains (Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Function, Role-Emotional and Mental Health) are derived and normalised to a scale of 0 to 100. The physical and mental component scores (PCS and MCS) are derived by multiplying each of these 8 scores by a constant, summing them and standardising against a population with a mean of 50, standard deviation of 10. A higher score represents a better quality of life. Mean changes from baseline score are presented as increases from baseline (defined as post-baseline minus baseline); larger changes indicate a better clinical condition. Mean refers to change in scores at Week 24. ANCOVA = analysis of covariance, BID = twice daily, DMARD = disease modifying antirheumatic drugs, PO = orally, QD = once daily
Time Frame: Baseline and 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | FOSTA 100 MG BID PO | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO | PLACEBO PO
Number analyzed (Participants) | 104 | 108 | 109
Units on a scale | 5 (8.3) | 4 (7.4) | 2 (6.2)
Statistical Analysis 1: Comparison: FOSTA 100 MG BID PO vs PLACEBO PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.009, ANCOVA; Improvement from baseline, including terms for baseline as a continuous covariate and treatment and pooled country as factors; Treatment difference = 2.60, 95% CI [0.65 to 4.56]
Statistical Analysis 2: Comparison: FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO vs PLACEBO PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.118, ANCOVA; [statistical method as in outcome 11, analysis 1]; Treatment difference = 1.53, 95% CI 2-sided [-0.39 to 3.44]

12. Secondary Outcome: SF-36 - Comparison of the Change in MCS From Baseline Between Fostamatinib and Placebo at Week 24
Description: SF-36: 36 item short form health survey, as a measure of health-related quality of life. The SF-36 scores for 8 sub-domains (Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Function, Role-Emotional and Mental Health) are derived and normalised to a scale of 0 to 100. The physical and mental component scores (PCS and MCS) are derived by multiplying each of these 8 scores by a constant, summing them and standardising against a population with a mean of 50, standard deviation of 10. A higher score represents a better quality of life. Mean changes from baseline score are presented as increases from baseline (defined as post-baseline minus baseline); larger changes indicate a better clinical condition. Mean refers to change in score at Week 24. ANCOVA = analysis of covariance, BID = twice daily, DMARD = disease modifying antirheumatic drugs, PO = orally, QD = once daily.
Time Frame: Baseline and 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | FOSTA 100 MG BID PO | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO | PLACEBO PO
Number analyzed (Participants) | 104 | 108 | 109
Units on a scale | 2 (8.6) | 2 (7.0) | 2 (7.3)
Statistical Analysis 1: Comparison: FOSTA 100 MG BID PO vs PLACEBO PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.487, ANCOVA; [statistical method as in outcome 11, analysis 1]; Treatment difference = 0.67, 95% CI [-1.23 to 2.58]
Statistical Analysis 2: Comparison: FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO vs PLACEBO PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.516, ANCOVA; [statistical method as in outcome 11, analysis 1]; Treatment difference = 0.62, 95% CI 2-sided [-1.26 to 2.51]

ADVERSE EVENTS:
Arm/Group | FOSTA 100 MG BID PO | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO | PLACEBO PO
Serious Adverse Events (participants affected / at risk) | 7/105 | 7/108 | 6/109
Other Adverse Events (participants affected / at risk) | 51/105 | 49/108 | 46/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FOSTA 100 MG BID PO (N=105) | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO (N=108) | PLACEBO PO (N=109)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
ARTERIOSCLEROSIS CORONARY ARTERY (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
CORONARY ARTERY OCCLUSION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
CROHN'S DISEASE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
GASTRIC ULCER (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1) | 1 (1) | 0 (0)
CHOLECYSTITIS (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
GASTROENTERITIS (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
GASTROENTERITIS BACTERIAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
HERPES PHARYNGITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
OROPHARYNGEAL CANDIDIASIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
TRANSIENT GLOBAL AMNESIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FOSTA 100 MG BID PO (N=105) | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO (N=108) | PLACEBO PO (N=109)
DIARRHOEA (Gastrointestinal disorders) | 21 (23) | 29 (31) | 7 (8)
FLATULENCE (Gastrointestinal disorders) | 6 (7) | 2 (2) | 4 (4)
NAUSEA (Gastrointestinal disorders) | 4 (5) | 7 (8) | 9 (9)
VOMITING (Gastrointestinal disorders) | 1 (1) | 6 (6) | 4 (4)
FATIGUE (General disorders) | 0 (0) | 0 (0) | 6 (6)
NASOPHARYNGITIS (Infections and infestations) | 6 (6) | 4 (5) | 4 (4)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 6 (7) | 2 (2) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 6 (6) | 0 (0) | 5 (5)
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 4 (5) | 6 (9) | 11 (11)
DIZZINESS (Nervous system disorders) | 7 (9) | 6 (6) | 2 (2)
HEADACHE (Nervous system disorders) | 8 (8) | 9 (9) | 11 (12)
HYPERTENSION (Vascular disorders) | 14 (15) | 15 (15) | 9 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No